CLINICAL TRIAL: NCT02925091
Title: Primary Antimicrobial Resistance Patterns of Austrian Helicobacter Pylori Clinical Isolates
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christoph Steininger, Assoc. Prof., Medical University of Vienna
Other Study IDs: MUVienna_Helicobacter
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Helicobacter pylori infects ~ 50% of the world's population and a quarter of the European population. H. pylori is responsible for a large proportion of gastric and duodenal ulcers and gastritis. Chronic infection with H. pylori is a risk factor for the development of stomach cancer and MALT (mucosa-associated lymphoid tissue) Lymphoma. The prospects of success for an antimicrobial eradication therapy is drastically reduced by the significant increase in antibiotic resistance in Austrian H. pylori isolates. The currently available data were obtained however from narrowly defined geographical regions and the clinical routine without information on patient selection. We suspect a considerable geographical variability of resistance patterns and a clinical bias for a preferential investigation of patients with unsuccessful, empirical eradication therapy. The objective of the proposed study is therefore an Austria-wide collection of data on H. pylori resistance in a prospective clinical study. The data thus collected will enable a significant improvement in current treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a diagnostic gastroscopy for the first time in their lives or had a diagnostic gastroscopy for any reason >10 years ago
* Older than 18 years of age
* Written informed consent

Exclusion Criteria:

* Previous H. pylori eradication therapies
* Antimicrobial treatment for other reasons than H. pylori eradication within 3 months prior to gastroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergoing a diagnostic gastroscopy for the first time in their lives or had a diagnostic gastroscopy for any reason >10 years ago
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Antimicrobial resistance of H. pylori isolate | 1 day (Once)

REFERENCES:
- [Derived] Bilgilier C, Stadlmann A, Makristathis A, Thannesberger J, Kastner MT, Knoflach P, Steiner P, Schoniger-Hekele M, Hogenauer C, Blesl A, Datz C, Huber-Schonauer U, Schofl R, Wewalka F, Puspok A, Mitrovits N, Leiner J, Tilg H, Effenberger M, Moser M, Siebert F, Hinterberger I, Wurzer H, Stupnicki T, Watzinger N, Gombotz G, Hubmann R, Klimpel S, Biowski-Frotz S, Schrutka-Kolbl C, Graziadei I, Ludwiczek O, Kundi M, Hirschl AM, Steininger C; Austrian Helicobacter Study Group of the Austrian Society of Gastroenterology and Hepatology. Prospective multicentre clinical study on inter- and intrapatient genetic variability for antimicrobial resistance of Helicobacter pylori. Clin Microbiol Infect. 2018 Mar;24(3):267-272. doi: 10.1016/j.cmi.2017.06.025. Epub 2017 Jun 29. PMID 28669844